CLINICAL TRIAL: NCT05564195
Title: Cognitive Trajectories After Surgery, a Clinical, Observational Feasibility Study
Acronym: POCOR
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Ulrica Nilsson, Professor, Karolinska Institutet
Other Study IDs: 2022-03593-01
Record Dates: First submitted 2022-09-02; First posted 2022-10-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing elective surgery with a duration of > 60 minutes: Participants included will be patients undergoing planned non-cardiac surgery with general anesthesia that are >60 years of age, have a Mini-mental state examination score of >24, are able to speak Swedish and does not suffer from uncorrected severe visual or auditory disorder, disease of the central nervous system, psychiatric diseases including alcoholism or drug dependence, current motor impairment in dominant hand, or colour-blindness.
  Interventions: Diagnostic Test: Postoperative cognitive function

INTERVENTIONS:
Diagnostic Test: Postoperative cognitive function — Digital cognitive tests - Mindmore-P, will be used to assess neurocognitive capacity and includes tests of verbal episodic memory, executive functions, visuospatial function and attention. The cognitive tests are self-administered on a touch screen tablet (10.1" 20-30 min Windows). The Mindmore-P is a web-application running on a full-screen Chrome browser. The test is administered by using a capacitive touchscreen with features that record detailed information such as timing, pauses, and lifting of finger from the touchscreen. Speech recognition is used in the screening of verbal memory and language.

SUMMARY:
Research problem and specific questions: Approximately 2.8 million surgeries are conducted yearly in Sweden and of these almost 50% are persons ≥ 60 years. Postoperative cognitive recovery is a concern for older persons. To date, there is no evidence for treating postoperative neurocognitive decline (POCD) and no assessment of cognitive function is routinely performed. The purpose is to is to test digital monitoring in clinical practice: I) test recruitment process and measure attrition rate; II) estimate the difference in main clinical outcomes (POCD) that will inform sample size calculations for the longitudinal observational mixed methods study, III) determine the usability and feasibility of digital monitoring. Participants: 50 patients ≥60 years undergoing inpatient surgery. Outcomes: depression, frailty, cognitive function, postoperative recovery and functional status .

DETAILED DESCRIPTION:
The aim is to evaluate the digital cognitive monitoring (Mindmore-P) in clinical practice by:

I) Test recruitment process and measure attrition rate. II) To establish whether it is possible to detect early signs of neurocognitive decline, using a digital postoperative cognitive screening tool i.e. Mindmore-P.

III) To investigate if there are any associations between choice of anesthetic drugs, delirium, duration of anesthesia, preoperative frailty, depression symptoms, postoperative delirium, physical function, and early postoperative recovery.

IV) Determine the usability and feasibility of Mindmore-P. V) Determine patients' experiences of early cognitive recovery in relation to signs of cognitive decline or no signs measured bythe four tests included in Mindmore-P

METHODS AND ANALYSIS Study design This is an observational feasibility study.

Participants included will be patients undergoing planned non-cardiac surgery with general anesthesia (n=50) at a hospital in Stockholm, Sweden. The sample size is based on the incidence of early cognitive decline at 1-2 weeks postoperatively of approximately 13-25%.

Inclusion criteria:

1. >60 years of age undergoing elective non-cardiac surgery with general anesthesia.
2. Duration of surgery >60 minutes
3. Mini-mental state examination (MMSE) score >24.

Exclusion criteria:

1. Unable to read and speak Swedish
2. Uncorrected severe visual or auditory disorder, disease of the central nervous system, psychiatric diseases including alcoholism or drug dependence, current motor impairment in dominant hand, or colour-blindness.

Recruitment At the patient's preoperative anaesthesia consultation, a research nurse will provide oral and written information about the study. The details of the study and its potential benefits as well as risks will be explained carefully to the patient. If the patient agrees to participate in the study, they will undergo a MMSE screening to examine if they are eligible for the study.

Outcomes, look below.

Analysis Descriptive statistics of demographic data will be presented with number, percentage, and mean (sd) or min-max, as appropriate. As recommended by Borchers et al review from 2021, mild POCD (1-2 standard deviation [sd]) and major POCD (>2 sd) will be specified for each test result and POCD is present if at least two tests indicates decline.

Usability and attrition rates will be presented with descriptive statistics. Preoperative depression (GDS), frailty (CFS), postoperative recovery (SwQoR), functional status (WHODAS) will be compared between the groups, using Kruskal Wallis ANOVA followed by Mann-Whitney U-test and a Bonferroni correction. To analyse intraindividual differences over time in cognitive performance, the same statistical tests will be used as well as multivariate logistic regression analysis. A p-value of <0.05 will be statistically significant in all analyses, Qualitative data will be analysed with thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* >60 years of age undergoing elective non-cardiac surgery with general anesthesia.
* Duration of surgery >60 minutes
* Mini-mental state examination score >24.

Exclusion Criteria:

* Mini-mental state examination, cut-off score of <23 indicating cognitive impairment
* Unable to read and speak Swedish
* Uncorrected severe visual or auditory disorder,
* Disease of the central nervous system
* Psychiatric diseases
* Alcoholism or drug dependence
* Current motor impairment in dominant hand
* Colour-blindness.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants included will be patients undergoing planned non-cardiac surgery with general anesthesia (n=50) at a hospital in Stockholm, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Recruitment process and attrition rate | Through study completion, an average of 8 months
  Number of possible participants vs. number of participants who accept to participate and number of participants who complete the study
Changes in postoperative cognitive function, part 1 | Before surgery and day 1 or 2, and 3 weeks after surgery
  Consortium to Establish a Registry for Alzheimer´s Disease (CERAD) A 10-word verbal learning test with 3 learning trials, a recall trial after ~7 min.
Changes in postoperative cognitive function, part 2 | Before surgery and day 1 or 2, and 3 weeks after surgery
  Trail Making Test (TMT- A & B), consisting of of 25 circles with letters or numbers on the screen.
  4. Symbol Digits Processing Test (SDPT).The test consist of nine symbol-digit pairings at the top of the screen, one symbol in the middle of the screen, and a number grid at the bottom of the screen.
Changes in postoperative cognitive function, part 3 | Before surgery and day 1 or 2, and 3 weeks after surgery
  Stroop Colour-Word Test (SCW). 24 words spelling out a the name of a colour which is printed in contrasting ink colours (e.g., the word "green" printed with red ink), and the participant is asked to tell the printed colour of the word rather than the word rather than the actual meaning of the word.
Changes in postoperative cognitive function, part 4 | Before surgery and day 1 or 2, and 3 weeks after surgery
  Symbol Digits Processing Test (SDPT).The test consist of nine symbol-digit pairings at the top of the screen, one symbol in the middle of the screen, and a number grid at the bottom of the screen.

SECONDARY OUTCOMES:
Frailty | Before surgery
  Clinical Frailty Scale, including 9-item ranging from 1 - very vital to 9 - terminally ill.
Signs of and changes in depression | Before surgery and 3 weeks after surgery
  Geriatric Depression Scale (GDS), consisting of 15 items to be answered with Yes or No. A score of 5 to 10 indicates probable depression and a score of more than 10 indicates definite depression.
Changes in functional capacity | Before surgery and 3 weeks after surgery
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS), thats consists of 12-item. Sum score ranges from 0-48, with increasing scores reflecting increasing disability
Changes in postoperative recovery | Before surgery and day 1 or 2, and 3 weeks after surgery
  Swedish version of Quality of Recovery, SwQoR, including 24 different postoperative symptoms to be rated on 11-point numerical scales from 0, "none of the time", to 10, "all of the time" Global score ranging from 0, "excellent quality of postoperative recovery," to 240, "extremely poor quality of recovery," with cutoff values of less than 31 at day 7 and less than 21 at day 14 indicating good recovery
Usability of Mindmore-P | 3 weeks after surgery
  System Usability Scale (SUS), consisting of 10 items to be answered on a 5-point scale from "strongly agree" to "strongly disagree".
Feasibility and patients' experiences of early postoperative cognitive recovery | One month after surgery
  Semi-structured, one-on-one interviews exploring patients' experiences of being assessed for cognitive performance and using Mindmore-P including assessment of facilitators and barriers, will be conducted. The participants will be asked to communicate freely on their experiences of their postoperative recovery.
Signs of and changes in postoperative delirium | After surgery twice a day on postoperative day 1-2
  Nursing Delirium Screening Scale NU-DESC, an observational five-item scale where symptoms delirium are rated from 0 to 2. A score of 2 or more indicates delirium

CONTACTS AND LOCATIONS:
Overall Officials: Ulrica Nilsson, Professor, Principal Investigator — Karolinska Insitutet
Locations (1):
- Ulrica Nilsson, Stockholm, Sweden

REFERENCES:
- [Derived] Amirpour A, Eckerblad J, Thorell A, Bergman L, Nilsson U. Usability and feasibility of a digital cognitive screening tool measuring older adults' early postoperative neurocognitive recovery: a protocol for a pilot study. BMJ Open. 2023 Jul 21;13(7):e070404. doi: 10.1136/bmjopen-2022-070404. PMID 37479514